CLINICAL TRIAL: NCT01546194
Title: A Survey of Patient's Attitudes Towards Consent For Clinical Research In Anesthesiology
Status: Completed | Type: Observational
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Glenn Murphy, Director, Cardiac Anesthesia and Clinical Research, Endeavor Health
Other Study IDs: EH09-533
Record Dates: First submitted 2012-02-28; First posted 2012-03-07 (Estimated); Results first posted 2015-09-25 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Informed Consent
Keywords: Informed consent; Perioperative period; Morning of surgery; Anesthesiology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Morning consent: Consent process consisting of information only provided on the morning of surgery
  Interventions: Other: Phone call explaining the research project
- Phone call and morning consent: Consent process consisting of information provided on the morning of surgery. In addition, a phone call on the day prior to surgery will be provided to subjects explaining that they will be approached about participation in a clinical research project
  Interventions: Other: Phone call explaining the research project

INTERVENTIONS:
Other: Phone call explaining the research project — A phone call on the day before surgery will be provided to subjects explaining the nature of the clinical trial

SUMMARY:
In most current academic anesthesia groups, it appears that consent for research is acquired on the day of surgery. This practice raises concerns because the hospital may be regarded as a coercive environment and there may be the possibility that the immediate preoperative environment prohibits adequate time for understanding the research project and making an informed decision about participation. However, this is often the only opportunity for anesthesiologists to obtain research consent. The aim of the present investigation is to utilize a survey study to determine if patients at Evanston Hospital are comfortable consenting for research on the day of surgery

DETAILED DESCRIPTION:
Patients participating in approved, minimal risk clinical research projects will be approached by the study investigators. Consent for clinical research will be obtained on the day of surgery in the ambulatory surgery unit. In addition, some patients will be contacted by telephone on the day prior to surgery to be informed that they will be approached about participation in a research project. If patients agree to participate in the clinical trial, they will be provided with a self-addressed envelope containing the survey and a brief cover letter. The research team member will explain the purpose of the survey (to determine patients' attitudes towards research consent on the day of surgery). Subjects will be requested to complete the survey within a week of the surgical procedure. Two days after surgery, the research team will provide a follow-up call to determine if there are any questions about completing the survey. Although patient names will not be identified on the survey packet, all surveys will be coded with the subjects study number for subsequent analysis.

Questions are designed to investigate six areas of potential concern relating to informed consent; comprehension, situation (privacy/time), obligation (pressure) motivation, compunction (regrets), and satisfaction. Subjects will reply using a 5-point scale from 1=strongly disagree to 5=strongly agree.

ELIGIBILITY:
Inclusion Criteria:

* Patients participating in approved, minimal risk clinical research projects will be approached by the study investigators

Exclusion Criteria:

* Inability to speak English
* Refusal to participate in the clinical research projects

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients participating in approved, minimal risk clinical research projects in the Department of Anesthesiology at NorthShore University HealthSystem will be approached by the study investigators.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn S. Murphy, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Morning Consent | Phone Call and Morning Consent
Started | 100 | 100
Completed | 64 | 65
Not Completed | 36 | 35

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Morning Consent | Phone Call and Morning Consent | Total
Number analyzed (Participants) | 64 | 65 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (10) | 56 (11) | 56 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 31 | 95
  Male | 0 | 34 | 34

OUTCOME MEASURES:

1. Primary Outcome: Overall Patient Satisfaction With the Same-day Consent Process-total Number of Questions Answered With a Score of 0 to 10 (on a 11-point Scale From 0=Strongly Disagree to 10=Strongly Agree).
Description: Subjects will reply using a 11-point scale from 0=strongly disagree to 10=strongly agree.
Time Frame: First postoperative day
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Morning Consent | Phone Call and Morning Consent
Number analyzed (Participants) | 64 | 65
units on a scale | 9.5 [3 to 10] | 10 [5 to 10]

ADVERSE EVENTS:
Time Frame: 1 week
Description: Patients followed for complications in hospital and after discharge in original studies. This was a survey
Arm/Group | Morning Consent | Phone Call and Morning Consent
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/65
Other Adverse Events (participants affected / at risk) | 0/64 | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes